# Title of Research Study: Comparison of normothermia maintenance between resistive blanket and forced air warming systems in renal transplant surgery

#### **Investigator Team Contact Information:**

For questions about research appointments, the research study, research results, or other concerns, call the study team at:

Investigator Name: Cole Bennett, MD Investigator Departmental Affiliation:

Anesthesiology

Phone Number: (612) 402-7900 Email Address: bennettc@umn.edu Phone Number: (612) 625-7116 Email Address: nelso377@umn.edu

Study Staff (if applicable): Candace Nelson

If your doctor is also the person responsible for this research study, please note that he is interested in both your clinical care and the conduct of this research study. You have the right to discuss this study with another person who is not part of the research team before deciding whether to participate in the research.

Supported By: This research is supported by University of Minnesota Department of Anesthesiology with staff time and effort. Also, the Hotdog U102 device has been donated by the manufacturer for the study.


TEMPLATE LAST REVISED: 12/16/2019

# **Key Information About This Research Study**

The following is a short summary to help you decide whether or not to be a part of this research study. More detailed information is listed later on in this form.

#### What is research?

Doctors and investigators are committed to your care and safety. There are important differences between research and treatment plans:

- The goal of research is to learn new things in order to help groups of people in the future. Investigators learn things by following the same plan with a number of participants, so they do not usually make changes to the plan for individual research participants. You, as an individual, may or may not be helped by volunteering for a research study.
- The goal of clinical care is to help you get better or to improve your quality of life. Doctors can make changes to your clinical care plan as needed.

Research and clinical care are often combined. One purpose of this informed consent document is to provide you clear information about the specific research activities of this study.

### Why am I being asked to take part in this research study?

We are asking you to take part in this research study because you are going to receive anesthesia for your kidney transplant. Patients receiving anesthesia can have the tendency to become hypothermic (to get cold) during the surgery. This can be due to a variety of reasons. The maintenance of normal body temperature is important for all patients undergoing anesthesia to maintain important body functions. To help patients maintain normal body temperature during the surgery, a warming device is used. This study will compare the effectiveness of a resistive blanket warming device to the standard of care forced air warming device.

### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### Why is this research being done?

The purpose of this research is to compare the effectiveness of resistive blanket warming to forced air warming in maintaining body temperature in patients undergoing anesthesia for a kidney transplant.

The forced air warming system, Bair Hugger Model 635, has a heater unit that blows air into an "air blanket" that inflates and circulates warm air throughout the blanket and exits through tiny holes on the side of the blanket that touches the patient. The warmed air, however, is only able to move over the skin surface in areas of the body that are immediately next to the blanket and which are not compressing the blanket (which would block airflow). This warming system is the standard care.


TEMPLATE LAST REVISED: 12/16/2019

The resistive blanket warming system, Hotdog U102, is equivalent to an operating-room-safe electric blanket. When plugged in, a semiconductor layer within the resistive blanket generates heat. The heat primarily warms the patient through direct skin contact, but also warms the air around the patient where there is no direct skin contact.

### How long will the research last?

We expect that you will be in this research study from the beginning of your surgery through one hour following your surgery.

### What will I need to do to participate?

You will be asked to give your consent to be in this research study. Once you provide consent, you will be randomized (like a flip of the coin) to either getting the Bair Hugger Model 635 forced air warming system or the Hotdog U102 resistive blanket warming system during your surgery.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

### Is there any way that being in this study could be bad for me?

Participating in this research does not pose any identifiable risks beyond those that are normally encountered with transplant surgery and anesthesia and temperature management. Thermal injury to the skin is listed as a risk for all warming systems that contact the skin (including both forced air and resistive blankets) but such events are exceedingly rare when the equipment is used as intended. We will use the devices according to the manufacturer's recommendations of operating the devices.

Researchers will take appropriate steps to protect any information they collect about you. However, there is a slight risk that information about you could be revealed inappropriately or accidentally.

### Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research.

### What happens if I do not want to be in this research?

You do not have to take part in this study. If you choose not to participate, you will receive normal anesthesia care practices.

# **Detailed Information About This Research Study**

The following is more detailed information about this study in addition to the information listed above.

### How many people will be studied?

We expect about 130 people here at the University of Minnesota will be in this research study.

### What happens if I say "Yes, I want to be in this research"?

If you agree to participate in this study, you will be given a signed copy of this document. You will undergo your 

TEMPLATE LAST REVISED: 12/16/2019

kidney transplant surgery as planned. Once you consent, you will be randomized (like a flip of the coin) to receive either the Hotdog U102 resistive blanket heating system or the Bair Hugger Model 635 warming system. Your body temperature will be monitored closely and data about the performance of the used warming system will be collected.

### What are my responsibilities if I take part in this research?

You will not have any additional responsibilities with this study. The study is completed one hour after your surgery.

# What happens if I say "Yes", but I change my mind later?

If you take part in this research study, and want to leave, you should tell us. Your choice not to be in this study will not negatively affect your right to any present or future medical care, or your present or future employment. If you stop being in the research, information about you that has already been collected may not be removed from the study database.

#### Can I be removed from the research?

Your physicians (either surgeon or anesthesiologist) may withdraw you from the study at any time without your approval if there are any concerns for your safety (whether related to the study or not).

### Will it cost me anything to participate in this research study?

Taking part in this research study will not lead to any costs to you.

# What happens to the information collected for the research, including my health information?

We try to limit the use and sharing of your information, including research study records, any medical records and any other information about you, to people who have a need for this information. But we cannot promise complete confidentiality.

#### **Overview**

If you participate in this study, your information, including your health information, will be used and shared for purposes of conducting this research. As described later in this Consent Form, your information may also be used and shared for publishing and presenting the research results, future research, and any optional elements of the research you agree to in this Consent Form, which may include creating audio and video recordings of you. If you sign this Consent Form, you are giving us permission to use and share your health information for these purposes, and if we are using your medical records, you are giving permission to any health care providers who are treating you to share your medical records with us.

#### What health information will be made available?

Health information about you to be used and shared for the research includes those items checked by the


TEMPLATE LAST REVISED: 12/16/2019

research team below:

☑ Your medical records, which may include records from hospital and clinic visits, emergency room visits, immunizations, medical history and physical exams, medications, images and imaging reports, progress notes, psychological tests, EEG/EKG/ECHO reports, lab and pathology reports, dental records and/or financial records. These records may be used and shared for as long as this research continues.

☑ Information collected as part of this research study, including research procedures, research visits, and any optional elements of the research you agree to, all as described in this Consent Form. This information might not be part of your medical record, and may include things like responses to surveys and questionnaires, and information collected during research visits described in this Consent Form.

#### What about more sensitive health information?

Some health information is so sensitive that it requires your specific permission. If this research study requires any of this sensitive information, the boxes below will be marked and you will be asked to initial to permit this information to be made available to the research team to use and share as described in this Consent Form.

| ☐ My drug & alcohol abuse, diagnosis & treatment records (initial) |
|--------------------------------------------------------------------|
| ☐ My HIV/AIDS testing records (initial) |
| ☐ My genetic testing records (initial) |
| ☐ My mental health diagnosis/treatment records (initial) |
| ☐ My sickle cell anemia records (initial) |

#### Who will access and use my health information?

If you agree to participate in this study, your information will be shared with:

- The University of Minnesota research team and any institutions or individuals collaborating on the research with us;
- Others at the University of Minnesota and M Health/Fairview who provide support for the research or who oversee research (such as the Institutional Review Board or IRB which is the committee that provides ethical and regulatory oversight of research at the University, systems administrators and other technical and/or administrative support personnel, compliance and audit professionals (Such as the Quality Assurance Program of the Human Research Protection Program (HRPP)), individuals involved in processing any compensation you may receive for your participation, and others);
- The research sponsor(s), any affiliates, partners or agents of the sponsor(s) involved in the research, organizations funding the research, and any affiliates, partners or agents of the funding organization(s) involved in the research;

 TEMPLATE LAST REVISED: 12/16/2019

- Organizations who provide accreditation and oversight for research and the research team, and others
  authorized by law to review the quality and safety of the research (such as U.S. government agencies
  like the Food and Drug Administration, the Office of Human Research Protections, the Office of Research
  Integrity, or government agencies in other countries); and
- Organizations that process any payments that may be made to you for participating in this study, and any other individuals or organizations specifically identified in this Consent Form.

#### Additional sharing of your information for mandatory reporting

If we learn about any of the following, we may be required or permitted by law or policy to report this information to authorities:

- Current or ongoing child or vulnerable adult abuse or neglect;
- Communicable, infectious or other diseases required to be reported under Minnesota's Reportable Disease Rule;
- Certain wounds or conditions required to be reported under other state or federal law; or
- Excessive use of alcohol or use of controlled substances for non-medical reasons during pregnancy.

#### How will my information be used in publications and presentations?

We may publish the results of this research in scientific, medical, academic or other journals or reports, or present the results at conferences. Information that makes it easy to identify you (such as your name and contact information, SSN and medical records number) will not be part of any publication or presentation. If you have an extremely unique or rare condition that is not shared by many others, it is possible that some people may be able to determine your identity even without these identifiers.

#### What will be done with my data when this study is over?

Your data will not be used for any future research after this study is complete.

Do I have to sign this Consent Form and give my permission to make my information, including my health information, available for use and sharing?

No, you do not have to sign this Consent Form. But if you do not sign, you will not be able to participate in this research study. Treatment available outside of the study, payment for such treatment, enrollment in health insurance plans and eligibility for benefits will not be impacted by your decision about signing this Consent Form.

Does my permission for making my health information available for use and sharing ever expire?

No, there is no expiration date.

May I cancel my permission for making my health information available for use and sharing?

Yes. You may cancel your permission at any time by writing to the researcher at the address on the first page of this Consent Form. If you cancel your permission, you will no longer be in the research study. You may also want 

TEMPLATE LAST REVISED: 12/16/2019

to ask someone on the research team in canceling will affect any research related medical treatment. If you cancel your permission, any health information about you that was already used and shared may continue to be used and shared for the research study and any optional elements of the study to which you agree in this Consent Form.

#### What happens to my health information after it is shared with others?

When we share your information with others as described in this Consent Form, privacy laws may no longer protect your information and there may be further sharing of your information.

#### Will I be able to look at my records?

It is possible that the research team may not allow you to see the information collected for this study. However, you may access any information placed in your medical records after the study is complete.

### Will anyone besides the study team be at my consent meeting?

You may be asked by the study team for your permission for an auditor to observe your consent meeting. Observing the consent meeting is one way that the University of Minnesota makes sure that your rights as a research participant are protected. The auditor is there to observe the consent meeting, which will be carried out by the people on the study team. The auditor will not document any personal (e.g. name, date of birth) or confidential information about you. The auditor will not observe your consent meeting without your permission ahead of time.

### Whom do I contact if I have questions, concerns or feedback about my experience?

This research has been reviewed and approved by an IRB within the Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 (Toll Free: 1-888-224-8636) or go to <a href="mailto:z.umn.edu/participants">z.umn.edu/participants</a>. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

### Will I have a chance to provide feedback after the study is over?

The HRPP may ask you to complete a survey that asks about your experience as a research participant. You do not have to complete the survey if you do not want to. If you do choose to complete the survey, your responses will be anonymous.

If you are not asked to complete a survey, but you would like to share feedback, please contact the study team or the HRPP. See the "Investigator Contact Information" of this form for study team contact information and "Whom do I contact if I have questions, concerns or feedback about my experience?" of this form for HRPP contact information.


TEMPLATE LAST REVISED: 12/16/2019

### What happens if I am injured while participating in this research?

In the event that this research activity results in an injury, treatment will be available, including first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner, to you or your insurance company. If you think that you have suffered a research related injury let the study physicians know right away.

### Will I be compensated for my participation?

No, you will not be compensated for your participation in this study.

| Your signature documents your permission to take part in signed document. | this research. You will be provided a copy of thi | S |
|---|---|---|
| Signature of Participant | Date | |
| Printed Name of Participant | | |
| Signature of Person Obtaining Consent | Date | |
| Printed Name of Person Obtaining Consent | <u></u> | |
| WITNESS STATEMENT: The participant was unable to read or sign this consent for | m because of the following reason: | |
| ☐ The participant is illiterate | | |
| ☐ The participant is visually impaired | | |
| $\square$ The participant is physically unable to sign the consent form. Please describe: | | |
| ☐ Other (please specify): | | |


TEMPLATE LAST REVISED: 12/16/2019

For the Consent of Non-English Speaking Participants when an Interpreter is Used:

# 

Version Date: V2, 02/23/2022

Printed Name of Individual